CLINICAL TRIAL: NCT03381443
Title: Participant Satisfaction With Two Different Summative Assessment Methods - a Mixed Method Questionnaire Study
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: ILS_assessment_2017/2018
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Assessment Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERC: all students assessed by the methods used by the European Resuscitation Council
  Interventions: Other: different assessments
- AHA: all students assessed by the methods used by the American Heart Association
  Interventions: Other: different assessments

INTERVENTIONS:
Other: different assessments — coded survey about NTS and assessment

SUMMARY:
Participants of Immediate Life Support and Advanced Life Support Courses, where two different summative assessment methods were used are asked about their satisfaction with the assessment method using a questionnaire. Both quantitative questions using an 11-point-Likert scale as well as open-ended qualitative questions will be asked. The primary aim of this study is to find out which variant of summative assessment is perceived by course participants as testing their leadership competency best, immediately after the comparison as well as 1 year later to identify any long-term effects on the students.

ELIGIBILITY:
Inclusion Criteria:

* All 5th and 6th year medical students at the University of Bern, Switzerland, study year 2017/2018 and 2018/2019

Exclusion Criteria:

* Refusal to participate

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All 5th and 6th year medical students at the University of Bern, Switzerland, study year 2017/2018 and 2018/2019
Sampling Method: Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction with summative assessment methods during Life Support Courses | directly after assessment and 1 year later
  evaluation of NTS assessed by assessment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, Prof., Study Chair — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No